CLINICAL TRIAL: NCT02627898
Title: Effect of Green Tea Extract Administration on Arterial Stiffness in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Green Tea Extract on Arterial Stiffness in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Fernando Grover Paez, PhD, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUCS-INTEC-MV-TEVE-001
Record Dates: First submitted 2015-12-03; First posted 2015-12-11 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Green tea extract; Arterial stiffness; PWVao
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Green tea extract (Experimental): Individuals with T2DM controlled with metformin or glibenclamide, or both; with no hypertension neither treated with insulim
  Interventions: Drug: green tea extract
- Placebo (Placebo Comparator): Individuals with T2DM controlled with metformin or glibenclamide, or both; with no hypertension neither treated with insulim
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: green tea extract — Green tea extract capsules, 400mg 1 time daily with the first bite of eat meal
  Other Names: Sunphenon 90LB
  Arms: Green tea extract
Drug: placebo — Placebo capsules, 400mg 1 time daily with the first bite of eat meal
  Other Names: Calcined magnesia
  Arms: Placebo

SUMMARY:
Type 2 diabetes mellitus (T2DM) has become the epidemic of the XXI century. This chronic disease is also highly prevalent and primarily associated with an increased cardiovascular mortality and morbidity due to micro and macrovascular complications, where its pathophysiological mechanism accelerates the formation of the atherosclerotic process, fundamental element associated with arterial stiffness. The importance of anticipating the presence of a cardiovascular event lies precisely in the early detection of subclinical changes in the elastic arteries identified by measuring the pulse wave velocity. Having adequate pharmacological or non-pharmacological interventions that impact precisely in the reduction of pulse wave velocity contributes to a reduction of cardiovascular morbidity and mortality associated with DM2. Among non-pharmacological therapies they have been studied the benefits attributed to the use of green tea infusion either encapsulated or extract have been associated mainly with anti-inflammatory and antioxidant effects. There are both experimental and clinical studies that have shown benefits of administration of green tea (extract or infusion), and administered by different routes at different dosages and for varying times. But it has been noted that not all studies with green tea meet appropriate to draw conclusions about its benefits to cardiovascular level. However, it is proposed that the use of green tea extract with a highest amount of catechins through a controlled clinical trial could be a potential therapeutic strategy for changing hemodynamic alterations and arterial stiffness favorably in this particular group of patients DM2.

DETAILED DESCRIPTION:
The objetive is to evaluate the effect of administration of Green tea exctract on arterial stiffness in individuals with T2DM. The investigators will conduct a double-blind trial, randomized, placebo control group, each group 12 male and female patients of 35-65 years of age with T2DM, with no hypertension or treated with insulins. Randomization will determine who will receive the intervention during 8 week trial (Green tea extract capsule, 400 mg 1 time daily with the first bite of each meal or approved placebo capsules), both groups also will continue with their usual treatment. The clinical findings and laboratory test include a metabolic profile and biosafety, wich will be baseline and at 8 weeks. Body weight, body fat, body mass index (BMI) and blood pressure will be determined during the inicial and final visit, likewise, hemodynamics parameters of arterial stiffness like the aortic pulse wave velocity (PWVao), central pulse pressure (PPao), aortic augmentation index (IAxao) and central systolic blood pressure (cSBP) by an oscillometric monitoring system via BPLab ®. Adverse events and adherence to treatment will be documented. The statistical analysis: Mann-Whitney U Test and Wilcoxon exact test. It is considered with significance at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM
* Fasting plasma glucose >126 and <250 mg/dl at the time security
* Metformin monotherapy or with glibenclamide added
* Written informed consent

Exclusion Criteria:

* Hypertention
* Treated with insulin
* Use of antioxidant suplements or products with caffeine
* Woman pregnant or breastfeeding
* Untreated tyroid disease
* Total colesterol >400mg/dl
* Triglycerides >400mg/dl
* Liver enzimes (alt and ast) more tan twice the normal range
* Glomerular filtration rate <60ml/min (Cockcroft-Gault)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Aortic Pulse Wave Velocity measured in meters / second, at 12 weeks | baseline and 12 weeks
  Before and after intervention with oscillometric monitoring system via BPLab

SECONDARY OUTCOMES:
Change from Baseline in aortic pulse pressure measured in mm / Hg at 12 weeks | baseline and 12 weeks
  Before and after intervention with oscillometric monitoring system via BPLab
Change from Baseline in aortic Augmentation index measured in percentage at 12 weeks | baseline and 12 weeks
  Before and after intervention with oscillometric monitoring system via BPLab
Change from Baseline in central systolic blood pressure measured in mm / Hg at 12 weeks | baseline and 12 weeks
  Before and after intervention with oscillometric monitoring system via BPLab

OTHER OUTCOMES:
Change from Baseline in Fasting plasma glucose measured in mg / dL at 12 weeks | baseline and 12 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Total cholesterol measured in mg / dL at 12 weeks | baseline and 12 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Triglycerids measured in mg / dL at 12 weeks | baseline and 12 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in High-density lipoprotein colesterol measured in mg / dL at 12 weeks | baseline and 12 weeks
  Before and after intervention by friedewall formula
Change from Baseline in Low-density lipoprotein colesterol measured in mg / dL at 12 weeks | baseline and 12 weeks
  Before and after intervention by friedewall formula
Change from Baseline in Alanine aminotransferase measured in IU / L at 12 weeks | baseline and 12 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Aspartate aminotransferase measured in IU / L at 12 weeks | baseline and 12 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Creatinine measured in mg / dL at 12 weeks | baseline and 12 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Peripheral systolic blood pressure measured in mg / dL at 12 weeks | baseline and 12 weeks
  Before and after intervention using a digital baumanometer
Change from Baseline in Peripheral diastolic blood pressure measured in mg / dL at 12 weeks | baseline and 12 weeks
  Before and after intervention using a digital baumanometer
Change from Baseline in Body and visceral fat measured in centimeters ^ 2 at 12 weeks | baseline and 12 weeks
  Before and after intervention using an impedance bascula, Dualscan HDS-2000

IPD SHARING:
Plan to Share IPD: No